CLINICAL TRIAL: NCT01108887
Title: Assessment of Adherence, Effectiveness & Convenience of Rebif® Treatment in Relapsing Multiple Sclerosis Patients Using RebiSmart™.
Brief Title: An Observational Study for the Assessment of Adherence, Effectiveness and Convenience of Rebif® Treatment in Relapsing Multiple Sclerosis Patients Using RebiSmart™.
Acronym: SMART
Status: Completed | Type: Observational
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A., Geneva (Industry)
Responsible Party: Sponsor
Other Study IDs: EMR 701068-526
Record Dates: First submitted 2010-04-21; First posted 2010-04-22 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2013-09

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: Multiple Sclerosis, Relapsing-Remitting; RebiSmart; Rebif; Interferon beta-1a
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
RebiSmart™ is a device with an electronic injection log to monitoring adherence to therapy. Therefore RebiSmart is a tool for administering Rebif in multi-dose cartridges that may improve patient satisfaction and adherence to therapy. The objectives of this study are to evaluate adherence, effectiveness and convenience of treatment in subjects with relapsing multiple sclerosis (RMS) using RebiSmart to self-inject Rebif in a multi-dose cartridge.

DETAILED DESCRIPTION:
This is an observational, international, multicenter study planned to be conducted in RMS subjects using the RebiSmart auto-injector at 300 sites in 15 countries across Europe. The participating countries are Austria, Belgium, Czech Republic, Denmark, Estonia, France, Germany, Hungary, Lithuania, Portugal, Slovakia, Sweden, Switzerland, the Netherlands and the United Kingdom. Subjects with RMS naïve to treatment or currently being treated with Rebif multi-dose injected by RebiSmart for no more than 6 weeks and meeting the eligibility criteria will receive Rebif 22 or 44 mcg subcutaneously three time a week. The dose of Rebif will be titrated during the initial four weeks of treatment. The planned observational period per subject is 12 months. The study visits comprises of: Baseline or Day 1 (Visit 1), Month 6 (Visit 2), and Month 12 (Visit 3).

OBJECTIVES

Primary objective:

* To assess adherence to treatment in subjects with RMS using RebiSmart to self-inject Rebif in a multi-dose cartridge

Secondary objectives:

* To assess effectiveness and convenience of treatment in subjects with RMS using RebiSmart to self-inject Rebif in a multi-dose cartridge.

ELIGIBILITY:
Inclusion Criteria:

* Males and female subjects between 18-65 years of age (only in Germany: Males and females between 12 - 65 years of age in order to follow national medical society guidelines)
* Female subjects must be neither pregnant nor breast-feeding and must lack child-bearing potential as defined by either: a) Post-menopausal or surgically sterile, or b) Using a highly effective method of contraception for the duration of the study. This is defined as a method that results in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, and includes for instance implants, injectables, combined oral contraceptives, intra-uterine device (IUD), sexual abstinence or vasectomised partner
* Subjects diagnosed with Relapsing MS according to the revised McDonald Criteria (2005)
* MS-treatment naïve subjects or subjects treated with Rebif multi-dose injected by RebiSmart for no longer than 6 weeks prior to Baseline visit
* Subjects that are able to self-inject with RebiSmart (in the opinion of the physician)
* Subjects with Expanded Disability Status Scale (EDSS) score < 6 (inclusive) at Baseline
* Signed informed consent (in countries where subject signature is not mandatory: subject must be given the patient information)

Exclusion Criteria:

* Subjects experiencing a relapse within 30 days before Baseline
* Subjects who have participated in other studies within 30 days before Baseline
* Subjects who received any MS therapy within 6 months prior to study enrolment (e.g., other disease modifying drugs: immunomodulatory, immunosuppressive agents or combination therapy) with the exception of Rebif multi-dose injected by RebiSmart
* Any visual or physical impairment that precludes the subject from self-injecting the treatment using the RebiSmart
* Pregnancy and breast-feeding
* Serious or acute heart disease such as uncontrolled cardiac dysrhythmias, uncontrolled angina pectoris, cardiomyopathy, or uncontrolled congestive heart failure
* Current or past (within the last 2 years) history of alcohol or drug abuse
* Have any contra-indications to treatment with interferon beta-1a according to Summary of Product Characteristics

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects with RMS naïve to treatment or currently being treated with Rebif multi-dose injected by RebiSmart for no more than 6 weeks
Sampling Method: Non-Probability Sample
Enrollment: 912 (Actual)
Dates: Start 2009-09; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Adherence to treatment | Baseline to 12 months of treatment
  Proportion of expected number of injections completed during 12 months of treatment as captured by RebiSmart.

SECONDARY OUTCOMES:
Effectiveness and convenience of treatment | Baseline to 12 months of treatment
  Overall evaluation of RebiSmart use based on Convenience Questionnaire; reasons for missed injections; proportion of subjects who prematurely terminated treatment and reasons why, proportion of subjects remaining disease-free, proportion of subjects relapse free; mean number of relapses
Safety of treatment | Baseline to 12 months
  Recording of adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Serono, a division of Merck KGaA, Darmstadt, Germany
Locations (1):
- Merck Serono Observational Site, Breda, Netherlands

REFERENCES:
- [Derived] Bayas A, Ouallet JC, Kallmann B, Hupperts R, Fulda U, Marhardt K; SMART study group. Adherence to, and effectiveness of, subcutaneous interferon beta-1a administered by RebiSmart(R) in patients with relapsing multiple sclerosis: results of the 1-year, observational SMART study. Expert Opin Drug Deliv. 2015 Aug;12(8):1239-50. doi: 10.1517/17425247.2015.1057567. Epub 2015 Jun 22. PMID 26098143